CLINICAL TRIAL: NCT03198962
Title: Use of Amphetamine-type Stimulants and Its Relationship With HIV Incidence and Antiretroviral Adherence Among Thai Men Who Have Sex With Men and Transgender Women
Brief Title: Use of Amphetamine-type Stimulants & Its Relationship With HIV Incidence and Antiretroviral Adherence Among MSM and TG
Status: Completed | Type: Observational
Sponsor: Thai Red Cross AIDS Research Centre (Other)
Collaborators: amfAR, The Foundation for AIDS Research (Other); TREAT Asia (Unknown)
Responsible Party: Sponsor
Other Study IDs: Amphetamine-type stimulants
Record Dates: First submitted 2017-06-22; First posted 2017-06-26 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2022-04

CONDITIONS: HIV Infections
Keywords: ATS, Thai MSM TG, Use of amphetamine-type stimulants, HIV, adherence
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Groups A: At each visit, a series of self-administered questionnaires will be used to collect demographic, sexual behavioral risk and drug use data. HIV testing, risk reduction counseling, condoms & lubricants will also be provided at these visits. Syphilis serology, Chlamydia trachomatis/Neisseria gonorrhea testing from anal and urethral compartments will be performed at baseline, month 6,12,18. HIV-negative participants will be actively offered to visit the clinic for pre-exposure prophylaxis (PrEP), post-exposure prophylaxis (PEP) or STI services and encouraged to visit the clinic outside of the scheduled visits for these services whenever they feel needed. Adherence to PrEP, PEP, STI treatment will be evaluated in those who are prescribed these medications. Among HIV seroconverters, drug use patterns will be longitudinally monitored prior to and after HIV diagnosis. HIV seroconverters at month 6 or month 12 will be transferred to groups C, D dependent on drug use history.
- Groups C: At each visit, a series of self-administered questionnaires will be used to collect demographic, behavioral risk and drug use data. In addition, data on adherence to antiretroviral therapy (ART) will be collected. Risk reduction counseling, adherence counseling, condoms & lubricants will also be provided at these visits. Syphilis serology, Chlamydia trachomatis/Neisseria gonorrhea testing from anal and urethral compartments will be performed at baseline, month 6,12,18.
- Group B: At each visit, a series of self-administered questionnaires will be used to collect demographic, sexual behavioral risk and drug use data. HIV testing, risk reduction counseling, condoms & lubricants will also be provided at these visits. Syphilis serology, Chlamydia trachomatis/Neisseria gonorrhea testing from anal and urethral compartments will be performed at baseline, month 6,12,18.
- Group D: At each visit, a series of self-administered questionnaires will be used to collect demographic, behavioral risk and drug use data. In addition, data on adherence to antiretroviral therapy (ART) will be collected. Risk reduction counseling, adherence counseling, condoms & lubricants will also be provided at these visits. Syphilis serology, Chlamydia trachomatis/Neisseria gonorrhea testing from anal and urethral compartments will be performed at baseline, month 6,12,18. HIV-positive participants, if they have not yet started ART, will be referred to preferred hospitals to receive ART regardless of CD4 count according to the 2014 National Guidelines. Drug use patterns will be longitudinally monitored prior to and after ART initiation.

SUMMARY:
There are two stages in the study. In Stage 1, 2000 Thai MSM, MSW and TGW/TGSW will be screened at the Thai Red Cross Anonymous Clinic (TRCAC) or Besides walk-in clients of TRCAC, potential participants could be referred to TRCAC by Rainbow Sky Association of Thailand (RSAT), Service Workers In Group (SWING) Foundation and Sisters Foundation. Each participant will complete a short standardized questionnaire on risk behavior, including use of amphetamine-type stimulants (ATS) and other drugs. HIV testing will be done following usual HIV testing and counseling (HTC) guidelines. Stage 1 will collect data on ATS use in the community. The results from stage 1 will also be used to stratify participants for inclusion in stage 2 of the study.

Participants from the screening will be invited to participate in stage 2 of the study, which is the longitudinal cohort study. Recruitment will be stratified by HIV status and ATS use as listed in to ensure an adequate number of ATS users for data analysis. Participants in stage 2 will follow-up every 6 months for 18 months.

DETAILED DESCRIPTION:
Stage 1 Stage one includes recruitment, the informed consent process, enrollment into the study, completion of the stage 1 questionnaire, and HIV counseling and testing. MSM/TG who present for routine HTC will be pre-screened for inclusion and exclusion criteria by the HTC counseling staff. MSM/TG who meet the inclusion criteria will be informed about the study and if interested will complete the informed consent process. After providing consent, participants will fill out the stage 1 questionnaire before receiving the HIV test result.

After the HIV test result is known to be positive or negative, the research staff will assign the participant to a study group (A,B,C,D) based on the HIV and ATS use status, as defined in section 3.2.3. If the study group has not yet filled to maximum size, then the participant will be offered participation in Stage 2 though another informed consent process. If the participant agrees, then the research staff will confirm contact information and will inform the participant that they will receive a reminder before the next visit in 6 months by their method of choice (telephone, SMS, email, Line, Facebook, etc).

If the study group has reached its maximum size, then the participant will be informed that their involvement in the study is finished and will be thanked for their contribution.

Stage 2 Stage 2 is the longitudinal follow-up of participants over 18 months. All study groups will follow the same schedule of follow-up visits one time every 6 months for 3 visits. At each visit, participants will complete a follow-up questionnaire and have a blood test. There will be no differences in procedures based on ATS use. Follow-up procedures will be divided by HIV status.

The four groups and sample sizes are:

1. Group A: HIV negative, non-ATS user (n=275)
2. Group B: HIV negative, ATS user (n=70)
3. Group C: HIV positive, non-ATS user (n=130)
4. Group D: HIV positive, ATS user (n=35)

ELIGIBILITY:
Stage 1

Inclusion Criteria:

* Age 18 years or above
* Born biological male
* Self-identifies as MSM or transgender woman
* Thai citizen
* Resident in Bangkok or surrounding suburb
* Had sex with a male partner at least once in the previous 12 months
* Consents to participate in the study

Exclusion Criteria:

* Unable to perform any study procedures, or unable to commit to attend all study visits.
* Has a serious medical, psychological, or substance use problem that, in the opinion of the study staff, would prevent appropriate participation or adequate follow-up in the trial

Criteria: Stage 2

Inclusion Criteria:

* Must meet all of the criteria in stage 1, plus:
* Completed HIV test with result determined to be positive or negative
* Agrees to return for follow-up visits with testing per protocol every 6 months for 18 months
* Consents to participate in the study

Exclusion Criteria:

* Indeterminate HIV test result

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population is Thai MSM or TGW who present for HIV counseling and testing at one of the participating sites.
Sampling Method: Non-Probability Sample
Enrollment: 510 (Actual)
Dates: Start 2016-11-15 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2023-02-16 (Actual)

PRIMARY OUTCOMES:
amphetamine-type stimulants (ATS) | 5 years
  The study of amphetamine-type stimulants (ATS) use among HIV-negative and HIV-positive Thai MSM, MSW, TGW and TGSW in Bangkok. Pattern of ATS use over the study period and by HIV status will be described along with its associated demographic and behavioral risk characteristics. The effect of ATS use on HIV and STI incidence among HIV-negative participants and ART adherence and virologic suppression among HIV-positive participants will also be studied.

CONTACTS AND LOCATIONS:
Overall Officials: Nittaya Phanuphak, MD, PhD, Principal Investigator — Thai Red Cross AIDS Research Centre (TRCARC)
Locations (1):
- The Thai Red Cross AIDS Research Centre, Bangkok, Thailand